CLINICAL TRIAL: NCT02862535
Title: A Phase 1b Study to Evaluate the Safety and Tolerability of Andecaliximab (GS-5745) as Monotherapy and in Combination With Anti-Cancer Agents in Japanese Subjects With Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Study to Evaluate the Safety and Tolerability of Andecaliximab as Monotherapy and in Combination With Anti-Cancer Agents in Japanese Participants With Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated due to sponsor's decision to not pursue further development of andecaliximab in oncology
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-296-1884
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Results first posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-11

CONDITIONS: Gastric Adenocarcinoma
MeSH Terms: interventions — andecaliximab; S 1 (combination); Cisplatin; Oxaliplatin; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort 1: ADX (Experimental): Participants will receive andecaliximab (ADX) 800 mg every 2 weeks on Days 1 and 15 of each 28-day treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
  Interventions: Drug: Andecaliximab
- Cohort 2: ADX + S-1 + Cisplatin (Experimental): Participants will receive ADX 800 mg every 2 weeks on Days 1 and 15 of each 28-day treatment cycle in combination with S-1 orally twice daily plus cisplatin chemotherapy (dosage and regimen will be based on participant condition, investigator discretion, institutional practice, and/or the in-country label) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
  Interventions: Drug: Andecaliximab; Drug: S-1; Drug: Cisplatin
- Cohort 3: ADX + S-1 + Oxaliplatin (Experimental): Participants will receive ADX 1200 mg every 3 weeks on Day 1 of each 21-day treatment cycle in combination with chemotherapy (S-1 80 mg/day to 120 mg/day according to the body surface area orally twice daily for first 14 days of 21 day cycle plus oxaliplatin 100 mg/m^2) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study.
  Interventions: Drug: Andecaliximab; Drug: S-1; Drug: Oxaliplatin
- Cohort 4: ADX + Nivolumab (Experimental): Participants will receive ADX 800 mg every 2 weeks followed by chemotherapy (nivolumab 3 mg/kg) on Days 1 and 15 of each 28-day treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
  Interventions: Drug: Andecaliximab; Drug: Nivolumab

INTERVENTIONS:
Drug: Andecaliximab — Administered via intravenous (IV) infusion (approximately 30 minutes)
  Other Names: GS-5745
Drug: S-1 — Administered orally
  Arms: Cohort 2: ADX + S-1 + Cisplatin; Cohort 3: ADX + S-1 + Oxaliplatin
Drug: Cisplatin — Administered via IV infusion on Day 8 of every 5 weeks
  Arms: Cohort 2: ADX + S-1 + Cisplatin
Drug: Oxaliplatin — Administered via IV infusion for over 2 hours on Day 1 of each 21-day cycle
  Arms: Cohort 3: ADX + S-1 + Oxaliplatin
Drug: Nivolumab — Administered via IV infusion (approximately 60 minutes) every 2 weeks
  Arms: Cohort 4: ADX + Nivolumab

SUMMARY:
The primary objective of this study is to characterize the safety and tolerability of andecaliximab as monotherapy and in combination with anti-cancer agents in Japanese participants with inoperable advanced or recurrent gastric or recurrent gastroesophageal junction (GEJ) adenocarcinoma.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have been born in Japan and must not have lived outside of Japan for a period > 1 year in the 5 years prior to Day 1
* Must be able to trace their maternal and paternal ancestry of parents and grandparents as ethnically Japanese
* Histologically confirmed inoperable advanced gastric adenocarcinoma (including adenocarcinoma of the GEJ) or relapsed gastric adenocarcinoma
* Cohorts 1, 2, and 3: Human Epidermal Growth Factor Receptor 2 (HER2)-negative tumor (primary tumor or metastatic lesion). Enrollment in Cohort 4 is not restricted by HER2 status (adults with HER2-positive, HER2-negative, or unknown HER2 status are eligible)
* Cohort 1: Prior antitumor therapy or cytotoxic chemotherapy is acceptable. Individuals who are not eligible to receive standard treatments should enroll on the study.
* Cohorts 2 and 3: Prior antitumor therapy or cytotoxic chemotherapy for metastatic disease is not acceptable. Individuals must be chemo-naive in the metastatic setting
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 1
* Adequate baseline organ function (within 28 days prior to Day 1)
* Coagulation: International Normalized Ratio (INR) ≤ 1.5 (unless receiving anticoagulation therapy)
* For females of childbearing potential, willingness to use a protocol-recommended method of contraception from the screening visit throughout the study treatment period and for defined periods following the last dose of andecaliximab and/or anti-cancer agent(s)
* For males of childbearing potential having intercourse with females of childbearing potential, willingness to use a protocol-recommended method of contraception from the start of andecaliximab, throughout the study treatment period, and for protocol defined periods following the last dose of andecaliximab and/or anti-cancer agent(s)
* Willingness to comply with scheduled visits, drug administration plan, imaging studies, laboratory tests, other study procedures, and study restrictions
* In addition to the applicable criteria above, participants in Cohort 4 must meet additional inclusion criteria to be eligible for participation in this study:

  * Measurable gastric or GEJ adenocarcinoma
  * Must have progressed on at least 1 prior systemic therapy or line of treatment for unresectable/metastatic disease.
  * Activated partial thromboplastin (aPTT) ≤ 1.5 times the upper limit of normal
  * Thyroid function tests should be within normal limits.

Key Exclusion Criteria:

* History or evidence of a clinically significant disorder, condition, or disease that, in the opinion of the investigator and medical monitor would pose a risk to participant safety or interfere with the study evaluations, procedures, or completion
* Pregnant or lactating. Enrollment of lactating females after discontinuation of breastfeeding is not acceptable.
* Individuals with known central nervous system (CNS) metastases, unless metastases are treated and stable and the individual does not require systemic steroids
* Radiotherapy within 28 days of Day 1
* Myocardial infarction, symptomatic congestive heart failure (New York Heart Association Classification > Class II), unstable angina, or serious uncontrolled cardiac arrhythmia within the last 6 months of Day 1
* History of major surgery within 28 days of Day 1
* Serious systemic fungal, bacterial, viral, or other infection that is not controlled or requires IV antibiotics
* Individuals known to be positive for human immunodeficiency virus (HIV), hepatitis C infection (per local standard diagnostic criteria), or acute or chronic hepatitis B infection (per local standard diagnostic criteria)
* In addition to the applicable criteria above, participants in Cohort 4 who meet any of the following exclusion criteria will not be enrolled in this study

  * Have received only neoadjuvant or adjuvant therapy for gastric adenocarcinoma
  * Prior treatment with anti-cytotoxic T-lymphocyte-associated protein 4 (anti-CTLA-4) agents, anti-programmed cell death protein 1 (anti PD-1) or anti-programmed cell death ligand 1 (anti-PD-L1) agents, anti-programmed cell death ligand 2 (anti-PD-L2) agents, anti-matrix metalloprotease (anti-MMP) agents, or other immunomodulatory therapies

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (3):
- Japan (3):
  - Nagoya
  - Osaka
  - Tokyo

REFERENCES:
- [Result] Yamaguchi K, Satoh T, Muro K, Takashima A, Ichimura T, et al. Phase 1b Study of Andecaliximab as Monotherapy and in Combination With Nivolumab in Japanese Patients With Gastric or GEJ Adenoracinoma [Poster L9]. Presented at ASCO GI 2019 Gastrointestinal Cancers Symposium: Jan 17-19, 2019, San Francisco, CA, USA.
- [Result] Muro K, Yamaguchi K, Satoh T, Kadowaki S, Ichimura T, et al. Phase 1b Study of Andecaliximab in Combination With S-1 + Platinum Chemotherapy in Japanese Patients With Advanced Gastric or GEJ Adenocarcinoma [Poster G3]. Presented at ASCO GI 2019 Gastrointestinal Cancers Symposium: Jan 17-19, 2019, San Francisco, CA, USA.
- [Result] Muro K, Satoh T, Yamaguchi K, Kadowaki S, Sakai D, et al. Phase 1b Study of Andecaliximab (ADX) as Monotherapy and in Combination With Nivolumab (nivo) in Japanese Subjects With Gastric or GEJ Adenocarcinoma. Presented at the Japanese Gastric Cancer Association: Feb 28, 2019.
- [Result] Satoh T, Yamaguchi K, Muro K, Sakai D, Ichimura T, et al. Phase 1b Study of Andecaliximab (GS-5745, ADX) in Combination With S-1 + Platinum Chemotherapy in Japanese Subjects With Advanced Gastric or GEJ Adenocarcinoma. Presented at the Japanese Gastric Cancer Association: Feb 28, 2019.
- [Derived] Ooki A, Satoh T, Muro K, Takashima A, Kadowaki S, Sakai D, Ichimura T, Mitani S, Kudo T, Chin K, Kitano S, Thai D, Zavodovskaya M, Liu J, Boku N, Yamaguchi K. A phase 1b study of andecaliximab in combination with S-1 plus platinum in Japanese patients with gastric adenocarcinoma. Sci Rep. 2022 Jun 30;12(1):11007. doi: 10.1038/s41598-022-13801-1. PMID 35773363
- [Derived] Yoshikawa AK, Yamaguchi K, Muro K, Takashima A, Ichimura T, Sakai D, Kadowaki S, Chin K, Kudo T, Mitani S, Kitano S, Thai D, Zavodovskaya M, Liu J, Boku N, Satoh T. Safety and tolerability of andecaliximab as monotherapy and in combination with an anti-PD-1 antibody in Japanese patients with gastric or gastroesophageal junction adenocarcinoma: a phase 1b study. J Immunother Cancer. 2022 Jan;10(1):e003518. doi: 10.1136/jitc-2021-003518. PMID 34992093

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Japan. The first participant was screened on 20 Sep 2016. The last study visit occurred on 25 Oct 2019.
Pre-assignment Details: 39 participants were screened.
Groups:
- Cohort 1: ADX: Participants received andecaliximab (ADX) 800 mg as monotherapy via intravenous (IV) infusion (approximately 30 minutes) every 2 weeks on Days 1 and 15 of each 28-day treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
- Cohort 2: ADX + S-1 + Cisplatin: Participants received ADX 800 mg via IV infusion (approximately 30 minutes) every 2 weeks on Days 1 and 15 of each 28-day treatment cycle in combination with chemotherapy (S-1 administered orally twice daily plus cisplatin administered via IV infusion on Day 8 of every 5 weeks) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug. Dose of S-1 and cisplatin was based upon participant condition, investigator discretion, institutional practice or in country label.
- Cohort 3: ADX + S-1 + Oxaliplatin: Participants received ADX 1200 mg via IV infusion (approximately 30 minutes) every 3 weeks on Day 1 of each 21-day treatment cycle in combination with chemotherapy (S-1 administered at 80 mg/day to 120 mg/day according to the body surface area orally twice daily for first 14 days of 21 day cycle plus oxaliplatin administered via IV infusion at 100 mg/m^2 over 2 hours on Day 1 of each 21-day cycle) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study.
- Cohort 4: ADX + Nivolumab: Participants received ADX 800 mg via IV infusion (approximately 30 minutes) every 2 weeks followed by chemotherapy (nivolumab 3 mg/kg via IV infusion [approximately 60 minutes] every 2 weeks) on Days 1 and 15 of each 28-day treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
Period: Overall Study
Arm/Group | Cohort 1: ADX | Cohort 2: ADX + S-1 + Cisplatin | Cohort 3: ADX + S-1 + Oxaliplatin | Cohort 4: ADX + Nivolumab
Started | 9 | 6 | 10 | 11
Completed | 0 | 0 | 0 | 0
Not Completed | 9 | 6 | 10 | 11
Not completed — Death | 7 | 3 | 2 | 5
Not completed — Study Terminated by Sponsor | 1 | 3 | 8 | 5
Not completed — Enrolled, not Treated | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who took at least 1 dose of study drug.
Groups:
- Cohort 1: ADX: Participants received ADX 800 mg as monotherapy via IV infusion (approximately 30 minutes) every 2 weeks on Days 1 and 15 of each 28-day treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
- Cohort 2: ADX+S-1+Cisplatin: Participants received ADX 800 mg via IV infusion (approximately 30 minutes) every 2 weeks on Days 1 and 15 of each 28-day treatment cycle in combination with chemotherapy (S-1 administered orally twice daily plus cisplatin administered via IV infusion on Day 8 of every 5 weeks) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug. Dose of S-1 and cisplatin was based upon participant condition, investigator discretion, institutional practice or in country label.
- Cohort 3: ADX+S-1+Oxaliplatin: Participants received ADX 1200 mg via IV infusion (approximately 30 minutes) every 3 weeks on Day 1 of each 21-day treatment cycle in combination with chemotherapy (S-1 administered at 80 mg/day to 120 mg/day according to the body surface area orally twice daily for first 14 days of 21 day cycle plus oxaliplatin administered via IV infusion at 100 mg/m^2 over 2 hours on Day 1 of each 21-day cycle) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study.
- Cohort 4: ADX+Nivolumab: Participants received ADX 800 mg via IV infusion (approximately 30 minutes) every 2 weeks followed by chemotherapy (nivolumab 3 mg/kg via IV infusion [approximately 60 minutes] every 2 weeks) on Days 1 and 15 of each 28-day treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: ADX | Cohort 2: ADX+S-1+Cisplatin | Cohort 3: ADX+S-1+Oxaliplatin | Cohort 4: ADX+Nivolumab | Total
Number analyzed (Participants) | 8 | 6 | 10 | 10 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (14.7) | 69 (7.9) | 56 (15.1) | 63 (11.8) | 61 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4 | 1 | 9
  Male | 5 | 5 | 6 | 9 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 6 | 10 | 10 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 8 | 6 | 10 | 10 | 34
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs are any AEs with an onset date of on or after the date that ADX and if applicable, nivolumab was first administered and no later than 30 days after permanent discontinuation of ADX, or if applicable, 5 months after permanent discontinuation of nivolumab (whichever is later).
Time Frame: First dose date up to 82.4 weeks plus 30 days (or if applicable, up to 5 months after permanent withdrawal of nivolumab)
Population: The Safety Analysis Set included all participants who took at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: ADX | Cohort 2: ADX + S-1 + Cisplatin | Cohort 3: ADX + S-1 + Oxaliplatin | Cohort 4: ADX + Nivolumab
Number analyzed (Participants) | 8 | 6 | 10 | 10
percentage of participants | 100.0 | 100.0 | 100.0 | 100.0

2. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least one toxicity grade from baseline. If the relevant baseline laboratory value was missing, then any abnormality of at least Grade 1 observed within the specified time frame (first dose date up to 82.4 weeks plus 30 days (or if applicable, up to 5 months after permanent withdrawal of nivolumab)) was considered treatment-emergent.Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 was used for assigning toxicity grades to laboratory results for analysis.
Time Frame: as for outcome 1
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: ADX | Cohort 2: ADX + S-1 + Cisplatin | Cohort 3: ADX + S-1 + Oxaliplatin | Cohort 4: ADX + Nivolumab
Number analyzed (Participants) | 8 | 6 | 10 | 10
percentage of participants
  Any Laboratory abnormalities: Hematology | 87.5 | 83.3 | 90.0 | 70.0
  Any Laboratory abnormalities: Chemistry | 100.0 | 100.0 | 100.0 | 80.0
  Any Laboratory abnormalities: Coagulation: number analyzed (Participants) | 7 | 6 | 10 | 10
  Any Laboratory abnormalities: Coagulation | 0 | 0 | 0 | 10.0

3. Secondary Outcome: Cohort 1: Plasma Concentration of Andecaliximab
Description: Plasma concentration is defined as the measured drug concentration. Blood samples were drawn at pre-dose and 30 (±15) minutes after infusion on Day 1 of Cycles 2, 3, 5; End of study (EOS) (3 years and 1 month); Cycle 1 only: 30 (±15) minutes after infusion on Day 1; anytime on Day 2, 4, and 8; pre-dose and 30 (±15) minutes post infusion on Day 15. The duration of each cycle for Cohort 1, 2, and 4 was 28 days and for Cohort 3 was 21 days. Infusion duration = 30 to 35 minutes.
  * min=minutes
  * D=Days
  * C=Cycle
Time Frame: Pre-dose and 30 (±15) min after infusion on C2D1, C3D1, C5D1; EOS (3 years and 1 month); C1 only: 30 (±15) min after infusion on D1; anytime on D2, D4 and D8; Pre-dose and 30 (±15) minutes post infusion on D15
Population: The Pharmacokinetic (PK) Analysis Set included all enrolled participants who took at least 1 dose of study drug and had at least 1 nonmissing postdose concentration value reported by the PK laboratory with available data were analyzed. Due to program discontinuation data were not collected for Cohorts 2, 3, and 4.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Cohort 1: ADX
Number analyzed (Participants) | 8
nanograms per milliliter
  30 minutes Postdose: Cycle 1 Day 1 | 262,625.0 (57410.64)
  Postdose: Cycle 1 Day 2 | 211,875.0 (56688.21)
  Postdose: Cycle 1 Day 4: number analyzed (Participants) | 7
  Postdose: Cycle 1 Day 4 | 133,100.0 (57485.39)
  Postdose: Cycle 1 Day 8 | 90100.0 (18127.25)
  Predose: Cycle 1 Day 15: number analyzed (Participants) | 7
  Predose: Cycle 1 Day 15 | 54800.0 (12011.66)
  30 minutes Postdose: Cycle 1 Day 15: number analyzed (Participants) | 7
  30 minutes Postdose: Cycle 1 Day 15 | 310,971.4 (128,365.39)
  Predose: Cycle 2 Day 1: number analyzed (Participants) | 3
  Predose: Cycle 2 Day 1 | 122,200.0 (52872.68)
  30 minutes Postdose: Cycle 2 Day 1: number analyzed (Participants) | 3
  30 minutes Postdose: Cycle 2 Day 1 | 458,666.7 (211,613.64)
  Predose: Cycle 3 Day 1: number analyzed (Participants) | 2
  Predose: Cycle 3 Day 1 | 158,000.0 (16970.56)
  30 minutes Postdose: Cycle 3 Day 1: number analyzed (Participants) | 2
  30 minutes Postdose: Cycle 3 Day 1 | 349,300.0 (402,626.60)
  Predose: Cycle 5 Day 1: number analyzed (Participants) | 2
  Predose: Cycle 5 Day 1 | 154,500.0 (6363.96)
  30 minutes Postdose: Cycle 5 Day 1: number analyzed (Participants) | 2
  30 minutes Postdose: Cycle 5 Day 1 | 510,500.0 (136,471.61)
  End of study: number analyzed (Participants) | 5
  End of study | 61960.0 (37635.40)

4. Secondary Outcome: PK Parameter: Cmax of Andecaliximab
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: Cycle 1 only: 30 (± 15) minutes after the end of infusion on Day 1; anytime on Days 2, 4, and 8; prior to dosing on Day 15 (Cycle length= 28 days) (infusion duration= 30 to 35 minutes)
Population: Participants in the PK Analysis Set were analyzed. Due to program discontinuation data were not collected for Cohorts 2, 3, and 4.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Cohort 1: ADX
Number analyzed (Participants) | 8
micrograms per milliliter | 264.0 (56.42)

5. Secondary Outcome: PK Parameter: AUClast of Andecaliximab
Description: AUClast is defined as the area under the concentration versus time curve to the last measurable concentration of drug from time zero to the last observable concentration.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours*micrograms per milliliter(h*μg/mL)
Arm/Group | Cohort 1: ADX
Number analyzed (Participants) | 8
hours*micrograms per milliliter(h*μg/mL) | 33500.2 (8397.01)

6. Secondary Outcome: PK Parameter: AUC0-336h of Andecaliximab
Description: AUC0-336h is defined as the area under the concentration versus time curve from time zero to time 336 hour.
Time Frame: as for outcome 4
Population: Participants in the PK Analysis Set with available data were analyzed. Due to program discontinuation data were not collected for Cohorts 2, 3, and 4.
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | Cohort 1: ADX
Number analyzed (Participants) | 7
h*μg/mL | 34341.9 (8697.66)

7. Secondary Outcome: Number of Participants With Positive Anti-Andecaliximab Antibodies
Time Frame: Pre-dose on Day 1 of Cycles 1, 2, 3, 5, 7 and every third cycle and anytime at EOT (82.4 weeks) and EOS visit (maximum: 3 years and 1 month) (Each Cycle= 28 days for Cohort 1, 2 and 4; 21 days for Cohort 3)
Population: The Immunogenicity Analysis Set included all participants who took at least 1 dose of study drug and had at least 1 nonmissing postdose antidrug antibody status reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ADX | Cohort 2: ADX + S-1 + Cisplatin | Cohort 3: ADX + S-1 + Oxaliplatin | Cohort 4: ADX + Nivolumab
Number analyzed (Participants) | 8 | 6 | 10 | 10
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to 82.4 weeks plus 30 days (or if applicable, up to 5 months after permanent withdrawal of nivolumab) All-Cause Mortality: From study start date up to study completion date (3 years and 1 month)
Description: The Safety Analysis Set included all participants who took at least 1 dose of study drug.
Arm/Group | Cohort 1: ADX | Cohort 2: ADX + S-1 + Cisplatin | Cohort 3: ADX + S-1 + Oxaliplatin | Cohort 4: ADX + Nivolumab
All-Cause Mortality (participants affected / at risk) | 7/8 | 3/6 | 2/10 | 5/10
Serious Adverse Events (participants affected / at risk) | 2/8 | 2/6 | 1/10 | 5/10
Other Adverse Events (participants affected / at risk) | 8/8 | 6/6 | 10/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: ADX (N=8) | Cohort 2: ADX + S-1 + Cisplatin (N=6) | Cohort 3: ADX + S-1 + Oxaliplatin (N=10) | Cohort 4: ADX + Nivolumab (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: ADX (N=8) | Cohort 2: ADX + S-1 + Cisplatin (N=6) | Cohort 3: ADX + S-1 + Oxaliplatin (N=10) | Cohort 4: ADX + Nivolumab (N=10)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Epidermolysis (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Blepharitis (Eye disorders) | 0 | 0 | 0 | 1
Conjunctivochalasis (Eye disorders) | 0 | 0 | 1 | 0
Dacryostenosis acquired (Eye disorders) | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anal inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 2 | 4 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 2 | 2
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 5 | 4 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 3 | 3 | 3
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Fatigue (General disorders) | 3 | 2 | 2 | 3
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 3 | 1 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1 | 1
Pyrexia (General disorders) | 2 | 2 | 1 | 2
Thirst (General disorders) | 0 | 0 | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Contrast media allergy (Immune system disorders) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 1
Enteritis infectious (Infections and infestations) | 1 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 2
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 2 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 1
Amylase increased (Investigations) | 0 | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 3 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 3 | 3 | 2
Platelet count decreased (Investigations) | 0 | 1 | 5 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 3 | 4 | 2
Decreased appetite (Metabolism and nutrition disorders) | 3 | 5 | 5 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 10 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 1
Vagus nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 3 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1
Vascular pain (Vascular disorders) | 0 | 0 | 3 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/35/NCT02862535/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/35/NCT02862535/SAP_001.pdf